CLINICAL TRIAL: NCT00006434
Title: Tumor Lysate Pulsed-Dendritic Cell Vaccines After High-Dose Chemotherapy for Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1694; M01RR000042 (NIH)
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Dendritic cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Biological: tumor-pulsed dendritic cells

SUMMARY:
When patients relapse after primary chemotherapy for Non-Hodgkin's lymphoma, they may be eligible to receive high-dose chemotherapy with autologous stem cell support. Unfortunately high-dose chemotherapy is curative in less than half the patients who receive it. This study is being conducted to determine the safety, side effects, and the ability to respond to an investigational vaccine that consists of tumor-pulsed dendritic cells given with an immune stimulating drug called interleukin-2. The patient must have a lymphomatous node accessible for excision to prepare the vaccine. Dendritic cells are immune cells that are obtained from the blood, and are important in the body's immune response to foreign substances. This study will examine the response of the immune system after three vaccinations (composed of dendritic cells, which have been exposed to dead fragments of lymphoma cells) given beginning three months after transplant. Vaccination may result in sensitizing the patient's dendritic cells to his lymphoma cells, potentially resulting in an immune response against the lymphoma. Twelve patients will be treated on study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, aggressive and/or intermediate grade NHL, B-cell and T-cell.
* In relapse after first-line conventional chemotherapy. Primary therapy should include a doxorubicin-based regimen.
* Patients must have disease sensitive to induction chemotherapy, radiation therapy, and/or radioimmunotherapy. Successful treatment of CNS or meningeal disease is allowed.
* Patients must have accessible tumor for biopsy or excision.
* Cumulative total doxorubicin: <500 mg/m2
* Performance score 0-2
* No prior pelvic RT
* Patients with a prior malignancy are eligible if they were treated for cure and have no evidence of active disease.
* Patients may not be taking immunosuppressive agents.
* Informed Consent; IRB approval

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States